CLINICAL TRIAL: NCT05350384
Title: An Unusual Association Between Pancreatic Cancer and Purtscher-like Retinopathy: Presentation of a Unique Case
Brief Title: An Unusual Association Between Pancreatic Cancer and Purtscher-like Retinopathy
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Eva Intagliata, researcher, University of Catania
Other Study IDs: UCatania666
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Purtscher Retinopathy; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methylprednisolone — 1 g. of methylprednisolone in saline solution 250 cc once a day for 5 days, and one eye drops of Diclofenac per eye 3 times a day for 30 days

SUMMARY:
AN UNUSUAL ASSOCIATION BETWEEN PANCREATIC CANCER AND PURTSCHER-LIKE RETINOPATHY

DETAILED DESCRIPTION:
Purtscher's retinopathy may cause sudden loss of vision of varying severity, secondary to head or chest injury. Its pathophysiology is unclear. Purtscher's-like retinopathy has more attenuated clinical and objective features and can be associated with many non-neoplastic pathologies.

Otherwise, an association of this kind of retinopathy with malignancies has been described once in the Literature (multiple myeloma). We present a case report on a unique association between pancreatic cancer and Purtscher-type retinopathy.

ELIGIBILITY:
Inclusion Criteria: NONE -

Exclusion Criteria: NONE

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No population, only one patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
funduscopic examination | at the onset of symptoms
  At the funduscopic examination the back of the eye showed large yellow spots and retinal hemorrhages in the superficial retina. In the early stages, fluorescein angiography showed hypofluorescence in the area of the yellow-white patches while the late stages showed hyperfluorescence

SECONDARY OUTCOMES:
abdominal CT-scan | at the onset of symptoms
  CT scan of the abdomen revealed a large mass in the tail of the pancreas with direct extension to the vessels of splenic hilum and splenic vein thrombosis. A secondary invasion of the gastric wall and left adrenal gland was also demonstrated. Percutaneous needle biopsy was performed and histopathology showed moderate to poorly differentiated mucinous pancreatic adenocarcinoma.

OTHER OUTCOMES:
Unusual association between Purtscher-like retinopathy and a malignant disease (pancreatic cancer) | at the diagnosis
  Ocular history and medical history were irrelevant.
Therapy | after 1 month from diagnosis
  An improvement of the macular edema and of the sight was reported after one-month administrating 1 g. of methylprednisolone in saline solution 250 cc once a day for 5 days, and one eye drops of Diclofenac per eye 3 times a day. The patient was not found fit for surgical treatment of his pancreatic cancer and therefore oncologic palliative medical treatment was performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Eva Intagliata, Catania, Italy

IPD SHARING:
Plan to Share IPD: No